CLINICAL TRIAL: NCT03112564
Title: Evaluation of the Effectiveness and Safety of Endotracheal Intubation for Inhalational Anesthesia Without the Use of Muscle Relaxants or Analgesics
Brief Title: Endotracheal Intubation Without Muscle Relaxants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Antonio Romero Berrocal, Anesthesiology and Critical Care, Puerta de Hierro University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUPH:PI:13/15
Record Dates: First submitted 2017-03-29; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Muscle Relaxation; Intubation Complication
Keywords: Endotracheal intubation; muscle relaxants; inhalational anesthesia
MeSH Terms: conditions — Muscle Hypotonia | interventions — cisatracurium; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sevoflurane 8% + Intravenous fentanyl (Other): Avoidance of rocuronium/cisatracurium
  Interventions: Other: Avoidance of rocuronium/cisatracurium; Drug: Sevoflurane 8% + Intravenous fentanyl

INTERVENTIONS:
Other: Avoidance of rocuronium/cisatracurium — Anesthesia induction was performed at tidal volume, avoiding the use of analgesics and/or muscle relaxants with FGF of 6 L/min. Induction time was shortened as the FGF was increased. Once 5% sevoflurane end-tidal volume was reached, ventilation with facial mask was maintained for three more minutes. The time lapsed until the loss of blink reflex was achieved and orotracheal tube (OTT) was placed, difficulties in OTT placement, sevoflurane end-tidal volume after OTT placement, complications related to OTT insertion (movement, coughing, rigidity, apnea), mean arterial pressure (MAP) variations were measured. No muscle relaxants were given during surgery.
Drug: Sevoflurane 8% + Intravenous fentanyl — Sevoflurane 8% + Intravenous fentanyl was the regimen used for induction and maintenance of anesthesia

SUMMARY:
Prospective study conducted between March 2013 and November 2014 at Hospital Universitario Puerta de Hierro-Majadahonda, in Madrid, Spain to identify complications and evaluate the efficacy of pure inhalational anesthesia induction to achieve endotracheal intubation without the use of muscle relaxant and analgesic drugs.

DETAILED DESCRIPTION:
This is a prospective study conducted between March 2013 and November 2014 at Hospital Universitario Puerta de Hierro-Majadahonda, in Madrid, Spain, with the previous approval by the institutional clinical research ethics committee. A total of 91 subjects who underwent general, gastrointestinal, orthopedic, urology and neurological surgery were randomly selected and provided written informed consent before any study-related procedures were performed.

The aim of this study was to identify complications and evaluate the efficacy of pure inhalational anesthesia induction to achieve endotracheal intubation without the use of muscle relaxant and analgesic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female patients
* Age ≥ 18 years
* ASA ≤ 3
* Able to provide informed consent

Exclusion Criteria:

* Subjects with left ventricle ejection fraction (LEVF) ≤ 35%
* History of ischemic heart disease in the last year
* History of malignant hyperthermia
* Presence of thoracic drain tubes
* Increased intracranial pressure (ICP) or brain tumors, undergoing neurophysiological monitoring
* Hemodynamic instability or likely to become unstable during induction of anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2013-03-01 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2014-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events during intubation | Time from anesthesia induction to 12 hours after the end of surgery
  Measurement of time lapsed from the loss of blink reflex after anesthesia induction and endotracheal tube placement. Number of patients with difficulty for intubation and number of patients with mean arterial pressure variations.

SECONDARY OUTCOMES:
Subject satisfaction following surgery | from the end of surgery until the discharge day up to 7 days
  subjects opinion regarding surgery satisfaction was collected
Post operative nausea and vomiting | first 12 hours after surgery
  record of nausea and/or vomiting events

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Romero Berrocal, MD,PhD, Principal Investigator — Hospital Universitario Puerta de Hierro, Madrid, Spain
Locations (1):
- Hospital Universitario Puerta de Hierro, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scheller MS, Zornow MH, Saidman LJ. Tracheal intubation without the use of muscle relaxants: a technique using propofol and varying doses of alfentanil. Anesth Analg. 1992 Nov;75(5):788-93. doi: 10.1213/00000539-199211000-00024. PMID 1416135
- [Background] Savarese JJ, Caldwell JE, Lien CA, Miller RD. Pharmacology of muscle relaxants and their antagonists. Anesthesia. 2000;5:412-90.
- [Background] Stevens JB, Wheatley L. Tracheal intubation in ambulatory surgery patients: using remifentanil and propofol without muscle relaxants. Anesth Analg. 1998 Jan;86(1):45-9. doi: 10.1097/00000539-199801000-00009. PMID 9428849
- [Background] Joo HS, Perks WJ. Sevoflurane versus propofol for anesthetic induction: a meta-analysis. Anesth Analg. 2000 Jul;91(1):213-9. doi: 10.1097/00000539-200007000-00040. PMID 10866915
- [Background] Trepanier CA, Brousseau C, Lacerte L. Myalgia in outpatient surgery: comparison of atracurium and succinylcholine. Can J Anaesth. 1988 May;35(3 ( Pt 1)):255-8. doi: 10.1007/BF03010619. PMID 3289770
- [Background] Kirkbride DA, Parker JL, Williams GD, Buggy DJ. Induction of anesthesia in the elderly ambulatory patient: a double-blinded comparison of propofol and sevoflurane. Anesth Analg. 2001 Nov;93(5):1185-7, table of contents. doi: 10.1097/00000539-200111000-00026. PMID 11682393
- [Background] Thwaites A, Edmends S, Smith I. Inhalation induction with sevoflurane: a double-blind comparison with propofol. Br J Anaesth. 1997 Apr;78(4):356-61. doi: 10.1093/bja/78.4.356. PMID 9135350
- [Background] Knaggs CL, Drummond GB. Randomized comparison of three methods of induction of anaesthesia with sevoflurane. Br J Anaesth. 2005 Aug;95(2):178-82. doi: 10.1093/bja/aei149. Epub 2005 Apr 29. PMID 15863438
- [Background] Topuz D, Postaci A, Sacan O, Yildiz N, Dikmen B. A comparison of sevoflurane induction versus propofol induction for laryngeal mask airway insertion in elderly patients. Saudi Med J. 2010 Oct;31(10):1124-9. PMID 20953528
- [Background] Walpole R, Logan M. Effect of sevoflurane concentration on inhalation induction of anaesthesia in the elderly. Br J Anaesth. 1999 Jan;82(1):20-4. doi: 10.1093/bja/82.1.20. PMID 10325830
- [Background] Vidal MA, Calderon E, Martinez E, Pernia A, Torres LM. [Comparison of 2 techniques for inhaled anesthetic induction with sevoflurane in coronary artery revascularization]. Rev Esp Anestesiol Reanim. 2006 Dec;53(10):639-42. Spanish. PMID 17302078
- [Background] Siddik-Sayyid SM, Aouad MT, Taha SK, Daaboul DG, Deeb PG, Massouh FM, Muallem MA, Baraka AS. A comparison of sevoflurane-propofol versus sevoflurane or propofol for laryngeal mask airway insertion in adults. Anesth Analg. 2005 Apr;100(4):1204-1209. doi: 10.1213/01.ANE.0000148166.29749.3B. PMID 15781547
- [Background] Bel Marcoval I, Gambus Cerrillo P. [Risk assessment, prophylaxis and treatment for postoperative nausea and vomiting]. Rev Esp Anestesiol Reanim. 2006 May;53(5):301-11. Spanish. PMID 16827070
- [Background] Philip BK, Lombard LL, Roaf ER, Drager LR, Calalang I, Philip JH. Comparison of vital capacity induction with sevoflurane to intravenous induction with propofol for adult ambulatory anesthesia. Anesth Analg. 1999 Sep;89(3):623-7. doi: 10.1097/00000539-199909000-00014. PMID 10475291